CLINICAL TRIAL: NCT05388942
Title: Virtual Reality Hypnosis Versus Inhaled Nitrous Oxide to Reduce Anterior Shoulder Dislocations: an Open Multicenter Randomized Controlled Trial
Brief Title: Virtual Reality Hypnosis Versus Inhaled Nitrous Oxide in Anterior Shoulder Dislocation Reduction: an Open Multicenter Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PT21134
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Shoulder Dislocation
Keywords: shoulder dislocation; virtual reality; hypnosis
MeSH Terms: conditions — Shoulder Dislocation | interventions — Nitrous Oxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality hypnosis (VRH) (Experimental)
  Interventions: Procedure: Virtual reality hypnosis
- Nitrous oxide (NO) (Active Comparator)
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Procedure: Virtual reality hypnosis — VRH offers predefined hypnosis sessions with no need of trained physician or nurse or caregiver mobilization. Consisting of a headset including headphones and a virtual reality screen, VRH allow patients to select a visual and sound environment (e.g.: tropical beach, space, underwater…) into which the hypnotic speech is delivered. That way, the patient's attention is distracted and muscular relaxation is obtained, a major relaxation factor. HRV is simple, quick, and presumably safe.
  Arms: Virtual reality hypnosis (VRH)
Drug: Nitrous oxide — inhalation of NO usually used to help with ASD reduction but inhaled NO has safety and maintenance issues.
  Arms: Nitrous oxide (NO)

SUMMARY:
Anterior shoulder dislocation (ASD) is a common situation in the emergency department (ED). Quick reductions lead to reduced mid and long term complications. No technique is superior to one another. Inhaled nitrous oxide can deal with pain reduction and anxiety but its efficacy is not optimal, with safety issues. Virtual reality hypnosis (VRH), by distracting patients from their pain, may lead to a better muscular relaxation and an easier ASD reduction.

Our first objective is to evaluate the clinical interest of VHR compared to nitrous oxide, in ASD reduction. Our second objective is to evaluate the safety of VRH in ASD reduction.

Patients over 18 years presenting an ASD < 24 hours, will be illegible for enrollment in an open multicenter randomized controlled trial, conducted in the Great East Region in France.

ELIGIBILITY:
Inclusion Criteria:

* patients of 18 years and older
* consulting the ED for a ASD < 24 hours
* with or without history of ASD
* with social insurance

Exclusion Criteria:

* non anterior shoulder dislocation
* shoulder or facial fracture or multiple trauma patient
* dementia, psychosis
* uncontrolled epilepsy
* visual or hearing issues
* claustrophobia
* vascular or nervous lesion of the dislocated arm
* contraindication with the use of inhaled nitrous oxide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-10-09 (Actual); Primary Completion 2023-10-09 (Estimated); Study Completion 2024-01-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of ASD procedure time | Day 0

SECONDARY OUTCOMES:
Achievement of the reduction of ASD procedure | Day 0
Per-procedure pain | Day 0
  Visual analogue scale
Passage time in the ED | Day 0
Patient satisfaction | Day 0
  Likert scale in 5 points
Adverse events when using HRV | Day 0
Adverse events when using inhaled NO | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France